CLINICAL TRIAL: NCT06972498
Title: A Prospective, Single-Arm, Multicenter Clinical Study on the Efficacy and Safety of Ivosimab Combined With Chemotherapy as Neoadjuvant Therapy in Patients With Resectable pMMR/MSS Colorectal Cancer Liver Metastases
Brief Title: A Prospective Multicenter Study: Ivosimab + Chemotherapy as Neoadjuvant for Resectable pMMR/MSS CRC Liver Mets
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-099
Record Dates: First submitted 2025-05-04; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer With Liver Metastasis
Keywords: Immunotherapy
MeSH Terms: interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Prospective, Single-Arm, Multicenter Clinical Study on the Efficacy and Safety of Ivosimab Combine (Experimental): Patients will receive ivosimab combined with the XELOX/FOLFOX regimen, followed by radical surgery 4-6 weeks after the last dose; adjuvant chemotherapy will continue for 3 months postoperatively.
  Interventions: Drug: Patients will receive ivosimab combined with the XELOX/FOLFOX regimen, followed by radical surgery 4-6 weeks after the last dose; adjuvant chemotherapy will continue for 3 months postoperatively.

INTERVENTIONS:
Drug: Patients will receive ivosimab combined with the XELOX/FOLFOX regimen, followed by radical surgery 4-6 weeks after the last dose; adjuvant chemotherapy will continue for 3 months postoperatively. — Patients will receive ivosimab combined with the XELOX/FOLFOX regimen, followed by radical surgery 4-6 weeks after the last dose; adjuvant chemotherapy will continue for 3 months postoperatively.

SUMMARY:
The population receiving ivosimab combined with chemotherapy for neoadjuvant treatment of colorectal cancer liver metastasis.

DETAILED DESCRIPTION:
The population receiving ivosimab combined with chemotherapy for neoadjuvant treatment of colorectal cancer liver metastasis

ELIGIBILITY:
Inclusion Criteria:

- Patients voluntarily join this study and sign the informed consent form (including consent for relevant tests on collected biological samples).

Male or female, aged ≥18 years and ≤75 years. Patients with pathologically or cytologically confirmed colorectal adenocarcinoma liver metastasis, and immunohistochemistry or genetic testing confirms pMMR/MSS.

Treatment-naive or relapsed colorectal cancer liver metastasis patients. For relapsed patients, the following must be met: no systemic antitumor therapy or radiotherapy within the past 1 year.

Primary tumor has been or can be radically resected.

Liver metastases are resectable and can achieve NED (no evidence of disease) status, meeting the following criteria:

Expected to achieve R0 resection through surgical resection and intraoperative ablation; Sufficient residual liver volume to preserve liver function; No distant metastases other than the liver. Planned for radical surgery after neoadjuvant therapy following MDT (multidisciplinary team) discussion.

At least 1 measurable lesion defined by RECIST v1.1 criteria. ECOG performance status 0-1. Expected survival ≥12 months. No concomitant diseases that increase surgical risk to an unacceptable level.

Organ functions meet the following requirements (no use of any blood components, colony-stimulating factors, or other corrective treatment drugs within 14 days before enrollment):

Absolute neutrophil count ≥1.5×10⁹/L; Platelets ≥100×10⁹/L; Hemoglobin ≥90 g/L; Serum albumin ≥35 g/L; Thyroid-stimulating hormone (TSH) ≤1×ULN; Serum bilirubin ≤1.5×ULN; ALT and AST ≤3×ULN; International normalized ratio (INR) ≤1.5 or prothrombin time (PT) ≤1.5×ULN; Serum creatinine ≤1.5×ULN. Non-surgically sterilized patients or women of childbearing potential must use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during and for 3 months after the study treatment period. Non-surgically sterilized women of childbearing potential must have a negative serum or urine HCG test within 72 hours before study enrollment, and must not be lactating. Male patients with partners of childbearing potential must use effective contraception during the trial and for 3 months after the last dose.

In addition to routine outpatient and inpatient recruitment, patients will also be recruited through 易拉宝 (pop-up displays) and WeChat official account promotions.

Exclusion Criteria:

- Presence of distant metastases other than the liver. Liver metastases have received prior antitumor therapy (chemotherapy, targeted therapy, immunotherapy, interventional therapy, etc.).

Liver metastases are unsuitable for surgical treatment. Residual toxicity from prior chemotherapy (excluding alopecia), such as grade ≥2 peripheral neuropathy.

Prior use of any therapy targeting T-cell costimulatory signaling pathways (e.g., anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4).

Active bleeding, ulcers, intestinal perforation, intestinal obstruction, or uncontrolled hypertension (uncontrollable by medication).

History of another primary malignancy within the past 3 years or concurrent malignancy (except cured basal cell carcinoma of the skin and cervical in situ carcinoma).

Active hepatitis B or hepatitis C infection. Active autoimmune disease or history of autoimmune disease (examples include but are not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism; vitiligo is permitted; asthma completely resolved in childhood without adult intervention is permitted; asthma requiring bronchodilator intervention is excluded).

Current use of immunosuppressants or systemic corticosteroid therapy for immunosuppression (dose >10 mg/day prednisone or equivalent) within 2 weeks prior to enrollment.

Hypertension uncontrolled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); uncontrolled cardiac symptoms or diseases, including:

1. NYHA class ≥2 heart failure;
2. unstable angina;
3. myocardial infarction within the past 1 year;
4. clinically significant supraventricular or ventricular arrhythmia requiring treatment/intervention;
5. QTc >450 ms (male) or QTc >470 ms (female). Coagulation abnormalities (INR >2.0, PT >16 seconds), bleeding diathesis, or current use of thrombolytic/anticoagulant therapy (prophylactic low-dose aspirin or low-molecular-weight heparin is permitted).

Arterial/venous thromboembolic events within 6 months prior to randomization (e.g., cerebrovascular accident [including transient ischemic attack, intracerebral hemorrhage, cerebral infarction], deep vein thrombosis, pulmonary embolism).

Known hereditary or acquired bleeding/thrombotic diathesis (e.g., hemophilia, coagulation disorders, thrombocytopenia).

Urinalysis showing proteinuria ≥ ++ confirmed by 24-hour urine protein >1.0 g. Active infection, unexplained fever ≥38.5°C within 7 days prior to first dose, or baseline white blood cell count >15×10⁹/L.

Congenital or acquired immunodeficiency (e.g., HIV infection). Systemic diseases such as cardiopulmonary insufficiency precluding tolerance of general anesthesia for partial nephrectomy or radical nephrectomy (note: likely a typo; original mentions "renal surgery," but context is colorectal cancer-should this be "hepatic surgery"?).

Other factors judged by the investigator to potentially affect study results or necessitate premature termination (e.g., alcohol/drug abuse, severe comorbidities requiring concurrent treatment [including mental illness], severe laboratory abnormalities, family/social factors impacting safety/compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 4months
  The objective response rate (ORR) in resectable pMMR/MSS colorectal cancer liver metastasis (CRLM) patients after neoadjuvant treatment with ivosimab combined with XELOX/FOLFOX.

IPD SHARING:
Plan to Share IPD: No
Patient Privacy and Confidentiality: Strict data protection regulations (e.g., GDPR, HIPAA) may prohibit sharing identifiable patient data, especially if anonymization is insufficient to mitigate risks.